CLINICAL TRIAL: NCT05241665
Title: A First in Human Study of the SpectraWAVE Imaging System
Brief Title: First in Human Study
Status: Completed | Type: Observational
Sponsor: SpectraWAVE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-01
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group 1
  Interventions: Device: SpectraWAVE Imaging System
- Group 2
  Interventions: Device: SpectraWAVE Imaging System

INTERVENTIONS:
Device: SpectraWAVE Imaging System — Coronary imaging

SUMMARY:
Investigational, prospective, multi-site, first in human, feasibility evaluation

ELIGIBILITY:
Group 1:

Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Patient with an indication for percutaneous coronary intervention (PCI) including:

   * Angina (stable or unstable),
   * Silent ischemia (a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or fractional flow reserve (FFR) ≤0.80 or iFR ≤0.89 must be present),
   * Non-ST-elevation myocardial infarction (NSTEMI), or
   * Recent ST-Segment Elevation Myocardial Infarction (STEMI) (>48 hours from initial presentation and stable).
3. Patients will undergo cardiac catheterization and possible or definite PCI.
4. Signed written informed consent.

Angiographic Inclusion Criteria:

1. The target lesion must be located in a native coronary artery with visually estimated reference vessel diameter of ≥2.25 mm to ≤5.2 mm and diameter stenosis of ≥50% but <100%.
2. Lesion length <40 mm.

Exclusion Criteria:

1. Serum creatinine ≥ 2.5 mg/dL Note: chronic dialysis dependent patients are eligible for enrolment regardless of creatinine.
2. STEMI within 48 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital.
3. PCI within 24 hours preceding the study procedure.
4. PCI of a lesion within the target vessel within 6 months prior to the study procedure.
5. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including an Intra-Aortic Balloon Pump, at time of procedure.
6. Mobitz II second degree or complete heart block.
7. Unstable ventricular arrhythmias
8. Pulmonary edema (defined as patient with shortness of breath, evidence of volume overload on physical exam, and crepitations on physical exam (>1/3 of lungs) or radiographic interstitial or alveolar pulmonary edema).
9. Subject is intubated.
10. Left ventricular ejection fraction (LVEF) ≤30% by the most recent imaging test within 3 months prior to procedure. If no LVEF test result within 3 months is available, it must be assessed by echocardiography, multiple gated acquisition (MUGA), magnetic resonance imaging (MRI), ventriculography (LV gram) or other method.
11. Severe valvular disease (e.g., severe mitral regurgitation or severe aortic stenosis)
12. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past 6 months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc.).
13. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.

    Note: femoral arterial disease does not exclude the patient if radial access may be used.
14. Presence of 1 or more co-morbidities which reduces life expectancy to less than 6 months or may interfere with protocol study processes.
15. Subject has known hypersensitivity or contraindication to radiocontrast dye that cannot be adequately pre-medicated.
16. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
17. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
18. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
19. Subject has a history of bleeding diathesis or coagulopathy or has had a significant gastro-intestinal or significant urinary bleed within the past 6 months.
20. Subject is currently participating in another investigational drug or device clinical study that has not yet completed its primary endpoint.
21. Women who are pregnant or breastfeeding
22. Women of childbearing potential unless a pregnancy test is negative within 1 week before study procedure.
23. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or impact the scientific soundness of the clinical investigation results.

    Angiographic Exclusion Criteria:
24. Left main diameter stenosis ≥30% or left main PCI planned.
25. Study target lesion in a bypass graft.
26. The target lesion is an ostial right coronary artery (RCA) stenosis.
27. Chronic total occlusion (Thrombolysis in Myocardial Infarction (TIMI) flow 0/1) study target lesion.
28. Bifurcation study lesion with a planned dual stent strategy.
29. In-stent restenosis study target lesion.
30. Any study lesion characteristic resulting in the expected inability to deliver the catheter to the lesion pre and post PCI (e.g., moderate or severe vessel calcification or tortuosity).
31. The target lesion contains more than a small amount of thrombus (as assessed angiographically) or is a stent thrombosis.

Group 2:

Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Patient must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia (ischemia in the absence of chest pain or other anginal equivalents), unstable angina, or acute myocardial infarction) suitable for PCI.
3. Patients undergoing a clinically indicated PCI procedure meeting 1 or more of the following criteria:

   A) High clinical risk, defined as medication-treated diabetes mellitus, AND/OR B) High angiographic-risk lesion(s), with at least 1 target lesion in each target vessel meeting at least 1 of the following criteria; i. Target lesion is the culprit lesion responsible for either:
   * NSTEMI, defined as a clinical syndrome consistent with an acute coronary syndrome and a minimum troponin of 1 ng/dL (may or may not have returned to normal), OR
   * STEMI >48 hours from the onset of ischemic symptoms ii. long or multiple lesions (defined as intended total stent length in any single target vessel ≥28 mm), Note: For a long target lesion, this would permit treatment by a single long stent or overlapping stents.

   Note: For up to 2 target lesions located in a single target vessel and treated with non-overlapping stents, they may be located in a continuous vessel or split up between a main vessel and a side branch.

   iii. bifurcation intended to be treated with 2 planned stents (i.e., in both the main branch and side branch), and where the planned side branch stent is ≥ 2.5 mm in diameter by angiographic visual estimation, iv. angiographic severe calcification (defined as angiographically visible calcification on both sides of the vessel wall in the absence of cardiac motion), v. chronic total occlusion (CTO) (enrollment in this case performed only after successful antegrade wire escalation crossing and pre-dilatation), vi. in-stent restenosis of diffuse or multi-focal pattern. Lesion must be at or within the existing stent margin(s) and have angiographically visually assessed DS ≥70% or DS ≥50% with non-invasive or invasive evidence of ischemia.
4. All target lesions must have a visually estimated or quantitatively assessed %DS of either ≥70%, or ≥50% plus 1 or more of the following: an abnormal functional test (e.g., FFR, instantaneous wave-free ratio (iFR), stress test) signifying ischemia in the distribution of the target lesion(s) or biomarker positive acute coronary syndrome (ACS) with plaque disruption or thrombus.

   Note: For purposes of study eligibility, a minimum troponin of 1 ng/dL at the time of screening will be considered biomarker positive.
5. No more than 2 target lesions requiring PCI are present in any single vessel, and no more than 2 target vessels are allowed. Thus, up to 4 target lesions per patient in a maximum of 2 target vessels are allowed, including branches.

   Note: A lesion is defined as any segment(s) of the coronary tree, no matter how long, which is planned to be covered with 1 contiguous length of stent, whether single or overlapped. A bifurcation counts as a single lesion even if the side branch is planned to be treated.

   Note: All lesions in a target vessel that are intended to be treated by PCI are designated as target lesions, and at least 1 target lesion in each target vessel must meet angiographic high-risk inclusion criteria summarized above in 3B). The only exception is for patients who qualify for the trial based on medication-treated diabetes, in which case no target lesion is required to meet angiographic high-risk inclusion criteria.
6. All target lesions intended to be treated by PCI in the target vessel are amenable to imaging guided PCI.

   Example: If a qualifying angiographic high-risk lesion is in the proximal LAD, and there is a second target lesion in the distal LAD which is a focal lesion not otherwise meeting high-risk criteria, both the proximal LAD and distal LAD lesions must be amenable to intravascular imaging (e.g., no excessive tortuosity or calcification precluding delivering the catheter), and each lesion must undergo imaging guided stenting. Otherwise, the vessel should be excluded.
7. Subject must provide written Informed Consent prior to any study related procedure.

   Angiographic Inclusion Criteria:
8. The target lesion must be located in a native coronary artery with visually estimated reference vessel diameter of ≥2.0 mm to ≤5.2 mm and diameter stenosis of ≥50% but <100%.

Exclusion Criteria:

1. STEMI <48 hours from the onset of ischemic symptoms
2. Serum creatinine ≥ 2.5 mg/dL Note: Chronic dialysis dependent patients are eligible for enrolment regardless of creatinine.
3. Hypotension, shock or need for mechanical support or intravenous vasopressors at the time the patient would be undergoing the index procedure.
4. Congestive Heart Failure (CHF) (Killip class ≥2 or New York Heart Association (NYHA) class ≥3)
5. LVEF ≤30% by the most recent imaging test within 3 months prior to procedure. If no LVEF test result within 3 months is available, it must be assessed by echocardiography, multiple gated acquisition (MUGA), magnetic resonance imaging (MRI), ventriculography (LV gram) or other method.
6. Unstable ventricular arrhythmias.
7. Inability to take Dual Antiplatelet Therapy (DAPT) (both aspirin and a P2Y12 inhibitor) for at least 30 days in the patient presenting with an ACS or in the patient presenting with stable coronary artery disease (CAD), unless the patient is also taking chronic oral anticoagulation in which case a shorter duration of DAPT may be prescribed per local standard of care.
8. Planned major cardiac or non-cardiac surgery within 30 days after the index procedure Note: Major surgery is any invasive operative procedure in which an extensive resection is performed, e.g., a body cavity is entered, organs are removed, or normal anatomy is altered.

   Note: Minor surgery is an operation on the superficial structures of the body or a manipulative procedure that does not involve a serious risk. Planned minor surgery is not excluded.
9. Prior PCI within the target vessel within 12 months Note: Prior PCI within the target vessel within 12 months is allowed for in-stent restenosis (target lesion is the prior PCI site) if no more than 1 layer of previously implanted stent is present.

   Note: In-stent restenosis involving 2 or more layers of stent implanted at any time prior to index procedure (i.e., an earlier episode of in-stent restenosis previously treated with a second stent) is excluded.
10. Any planned PCI within the target vessel(s) within 30 days after the study procedure, other than a planned staged intervention in a second target vessel.

    Note: Planned staged interventions must be noted at the time of enrollment, and the decision to stage may be modified within 24 hours of completion of the index PCI.

    Note: PCI in non-target vessels is permitted >48 hours after the index procedure.
11. Any prior PCI in a non-target vessel within 24 hours before the study procedure, or within previous 30 days if unsuccessful or complicated.

    Note: Patients requiring non-target vessel PCI may be enrolled and the non-target vessel(s) may be treated in the same index procedure as the enrolled lesions (in all cases prior to enrollment), as long as treatment of the lesion(s) in the non-target vessel is successful and uncomplicated.

    Successful and uncomplicated definition for non-target vessel treatment during the index procedure: Angiographic diameter stenosis <10% for all treated non-target lesions, with TIMI III flow in this vessel, without final dissection ≥ National Heart, Lung, and Blood Institute (NHLBI) type B, perforation anytime during the procedure, prolonged chest pain (>5 minutes) or prolonged ST-segment elevation or depression (>5 minutes), or cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation).
12. Subject has known hypersensitivity or contraindication to radiocontrast dye that cannot be adequately pre-medicated.
13. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
14. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
15. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
16. Subject has a history of bleeding diathesis or coagulopathy or has had a significant gastro-intestinal or significant urinary bleed within the past 6 months.
17. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past 6 months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc.).
18. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.

    Note: femoral arterial disease does not exclude the patient if radial access may be used.
19. Subject has life expectancy <6 months for any non-cardiac cause.
20. Subject is currently participating in another investigational drug or device clinical study that has not yet completed its primary endpoint.
21. Women who are pregnant or breastfeeding
22. Women of childbearing potential unless a pregnancy test is negative within 1 week before procedure.
23. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or impact the scientific soundness of the clinical investigation results.

    Angiographic Exclusion Criteria:
24. Severe vessel tortuosity or calcification in a target vessel such that it is unlikely that the imaging catheter can be delivered.

    Note: severe vessel calcification is allowed if it is expected that the catheter can be delivered at baseline or after vessel preparation with balloon pre-dilatation or atherectomy.
25. The target vessel has a lesion with diameter stenosis (DS) ≥ 50% that is not planned for treatment at the time of index procedure.
26. The target lesion is in a bypass graft conduit. Note: A native coronary artery may be enrolled if a prior bypass graft conduit to the vessel is totally occluded, but not if it is patent.
27. The target lesion is an ostial RCA or ostial Left Main stenosis.
28. The target lesion contains more than a small amount of thrombus (as assessed angiographically) or is a stent thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects who are scheduled for coronary angiography and are candidates for percutaneous coronary interventional procedures.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Feasibility Evaluation | From informed consent to hospital discharge after the SpectraWAVE Imaging System procedure, an average of less than one day.
  The primary endpoint is the feasibility evaluation of the SpectraWAVE Imaging System to successfully image the native coronary artery as measured by questionnaire.

SECONDARY OUTCOMES:
Safety Evaluation | From informed consent to 30-Day Follow-Up Visit after the SpectraWAVE Imaging System procedure.
  The secondary endpoint will be the assessment of any adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Angiografia De Occidente S.A, Cali, Colombia

IPD SHARING:
Plan to Share IPD: No